CLINICAL TRIAL: NCT01474057
Title: Online Early Resilience Intervention for Combat-Related PTSD in Military Primary Healthcare Settings: A Randomized Trial of "DESTRESS-PC"
Brief Title: DElivery of Self Training and Education for Stressful Situations-Primary Care Version
Acronym: DESTRESS-PC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Charles Engel, Dir., Deployment Health Clinical Center, WRNMMC; Associate Professor, psychiatry, USUHS, Uniformed Services University of the Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: W81XWH-07-2-0006; 1R34MH078874-01 (NIH)
Record Dates: First submitted 2010-03-26; First posted 2011-11-17 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Posttraumatic Stress Disorder (PTSD)
Keywords: PTSD; combat trauma; telemedicine; primary care interventions; CBT; self-managed treatment; web-based intervention; internet treatment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DESTRESS-PC (Experimental): A brief, nurse-assisted, Internet-based online self-management tool for PTSD (DESTRESS-PC), based on empirically valid cognitive-behavioral therapy (CBT) strategies and designed for implementation in a primary care setting. DESTRESS-PC stands for DElivery of Self-TRaining and Education for Stressful Situations for Primary Care.
  Interventions: Behavioral: DESTRESS-PC
- OUC (Active Comparator): Optimized Usual Care (OUC) for PTSD--usual PTSD treatment offered within the primary care setting, optimized by training PC providers in PTSD identification and treatment and providing basic care management including phone check-ins to monitor symptoms and feedback to providers.
  Interventions: Other: Optimized Usual Primary Care PTSD treatment

INTERVENTIONS:
Behavioral: DESTRESS-PC — An online nurse-assisted, self-management intervention designed for primary care treatment of war-related PTSD, this intervention will consist of 3 weekly logins to a secure website for a period of 6 weeks. A "DESTRESS Nurse" will train the participant to use the website and will monitor their progress and report key information back to the primary care physician.
  Arms: DESTRESS-PC
Other: Optimized Usual Primary Care PTSD treatment — Participants receive usual Primary Care treatment that is administered by the primary care physician; the DESTRESS Nurse monitors the participants' progress throughout the study.
  Arms: OUC

SUMMARY:
This study will compare a cognitive-behavioral online self-management intervention designed for primary care treatment of war-related PTSD to a control intervention, "optimized usual primary care PTSD treatment". Patients with PTSD will be trained to use the online PTSD treatment website and asked to do so three times per week for six weeks. They will have phone and email access to a nurse trained to assist them in their treatment program. Three scheduled phone check-ins during the six week treatment period will provide ongoing contact with patients during treatment. The investigators will assess PTSD symptoms, depression, anxiety and somatic symptoms, physical health status and occupational functioning on three occasions: before the intervention, at the end of the treatment period, and six weeks after the end of treatment.

DETAILED DESCRIPTION:
The study is a multi-site trial evaluating the efficacy of DESTRESS-PC (DElivery of Self-TRaining and Education for Stressful Situations, primary care version), a brief, web-based self-management intervention for PTSD designed for delivery in primary care. Participants randomized to DESTRESS-PC log on to a secure website for self-CBT 3 times per week for 6 weeks and receive RN nurse care manager ("DESTRESS Nurse") contact every two weeks. DESTRESS Nurses introduce the approach, monitor, answer questions, and insure primary care provider collaboration. The control intervention is optimized usual primary care. Blinded raters assess PTSD symptoms, depression, anxiety, somatic symptoms, physical health status, and occupational functioning at four timepoints. All study participants receive RN care management and are under the care of a primary care provider trained in evidence-based PTSD treatment who receives status reports from the DESTRESS nurse to include baseline psychiatric status.

ELIGIBILITY:
Inclusion Criteria:

* Referred by a primary care providers in a participating primary care clinic.
* Deployed to either Operation Iraqi Freedom or Enduring Freedom.
* War-related trauma while deployed (may include military sexual trauma).
* Current PTSD as addressed by the CAPS interview.
* Reports routine access to computer, internet, and email.
* Successfully uses Internet to coordinate baseline assessment appointment.
* Provides research informed consent using local IRB-approved form.
* Plans continued care at the enrolling primary care clinic for at least 4 months.

Exclusion Criteria:

* Actively engaged in specialty mental health care in the previous two months.
* Failed specialty mental health treatment for PTSD or associated condition.
* Acute psychosis, psychotic episode, or psychotic disorder diagnosis within the past two years.
* Active substance dependence disorder in the past year.
* Active suicidal or violent ideation within the past two months.
* Currently on an antipsychotic or mood-stabilizing agent.
* Unstable administration schedule or dosing of any antidepressant, anxiolytic, or sedative-hypnotic (i.e., will exclude for any related medication changes in the two-months prior to randomization).
* Acute or unstable physical illness.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2008-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
PTSD Checklist (PCL) | Baseline and 6 weeks, 12 weeks, and 18 weeks post randomization
  Symptoms of PTSD were assessed using the PTSD Checklist-Military Version (PCL). The PCL is a self-report measure developed for measuring PTSD symptom severity and for estimating PTSD caseness when administration of a structured clinical interview is not feasible. Respondents rate PCL items on a 5-point scale ('not at all' through "extremely') to indicate the degree to which they have been bothered by each of 17 PTSD symptoms during the past month. Possible PCL scores range from 17 to 85.

SECONDARY OUTCOMES:
PRIME-MD PHQ | baseline and 6 weeks,12 weeks, and 18 weeks post randomization
  The PHQ is a brief self-report assessment of common mental disorders developed specifically for primary care. PHQ allows brief provisional primary care diagnoses of several disorders including major depression, panic disorder, other anxiety disorder, and multi-somatoform disorder. We used the PHQ for baseline and follow-up assessments of depression, anxiety (panic and generalized anxiety), and somatic symptom severity, assessments with excellent correspondence to DSM-IV diagnostic criteria.
Medical Outcomes Study Short Form-36 (SF-36) | baseline, 6 wks, 12 wks, and 18wks
  The SF-36 is a widely used measure of health related quality of life with established reliability and validity. The SF-36 was used to describe the study sample, compare functional status of the intervention groups at baseline, and assess change in functional over the course of the study.
Attitude Regarding Mental Health Treatments | baseline, 6 weeks, 12 weeks, and 18 weeks
  We used two questions from Hoge and colleagues (2004): 'I don't trust mental health professionals,' and 'Mental health care doesn't work.' Both questions are rated using a five-point Likert-type scale. We also used two questions that rate attitudes regarding psychotherapy treatment ('Psychotherapy patients are wasting money,' and 'Therapy can help an individual'). The latter two questions, rated on the same 5-point scale, were part of a longer measure used to evaluate stigma in primary care patients with anxiety disorders.
World Health Organization Health and Performance Questionnaire (HPQ). | baseline, 6 weeks, 12 weeks, and 18 weeks
  The HPQ is an assessment instrument to estimate the costs of workplace health problems using a self-report instrument. Specific areas assessed include job performance, absenteeism, and work related critical incidents.

CONTACTS AND LOCATIONS:
Overall Officials: Charles C. Engel, M.D., M.P.H., Principal Investigator — Uniformed Services University of the Health Sciences
Locations (4):
- United States (4):
  - Savannah Primary Care Clinic (Charleston VA), Savannah, Georgia
  - Department of Veterans Affairs, Boston, Boston, Massachusetts
  - Ralph H. Johnson VA Medical Center/Goose Creek Primary Care Clinic (Charleston VA), Charleston, South Carolina
  - Womack Army Medical Center, Fort Bragg, South Carolina

REFERENCES:
- [Background] Litz BT, Engel CC, Bryant RA, Papa A. A randomized, controlled proof-of-concept trial of an Internet-based, therapist-assisted self-management treatment for posttraumatic stress disorder. Am J Psychiatry. 2007 Nov;164(11):1676-83. doi: 10.1176/appi.ajp.2007.06122057. PMID 17974932
- [Background] Litz, BT, Williams, L, Wang, J, Bryant, R, and Engel, CC. A Therapist-Assisted Internet Self-Help Program for Traumatic Stress. Professional Psychology: Research and Practice 35(6):628-634, 2004.
- [Derived] Simon N, Robertson L, Lewis C, Roberts NP, Bethell A, Dawson S, Bisson JI. Internet-based cognitive and behavioural therapies for post-traumatic stress disorder (PTSD) in adults. Cochrane Database Syst Rev. 2021 May 20;5(5):CD011710. doi: 10.1002/14651858.CD011710.pub3. PMID 34015141